CLINICAL TRIAL: NCT05487378
Title: Randomised Investigation to Evaluate Phe Fluctuation in PKU Patients Treated With PKU GOLIKE Versus Standard Amino Acid Protein Substitute.
Brief Title: Evaluation of Phe Fluctuation in PKU Pts Treated With PKU GOLIKE Versus Standard Amino Acid Protein Substitute.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: APR Applied Pharma Research s.a. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: GLK-UK-2021
Record Dates: First submitted 2022-06-17; First posted 2022-08-04 (Actual); Results first posted 2025-06-08 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2023-10

CONDITIONS: Phenylketonurias
MeSH Terms: conditions — Phenylketonurias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1st PKU GOLIKE 2nd AA protein substitute (Other): 7 days with usual protein substitute and PKU GOLIKE as their last dose of protein substitute for the day (at least one sachet with15g PE) in an amount equivalent to their usual protein substitute PE followed by a 2-week washout period on their usual protein substitute, and then 7 days with AA protein substitute for all daily doses.
  Interventions: Dietary Supplement: PKU GOLIKE
- 1st AA protein substitute 2nd PKU GOLIKE (Other): 7 days with AA protein substitute for all daily doses followed by a 2-week washout period on their usual protein substitute, and then 7 days with usual protein substitute and PKU GOLIKE as their last dose of protein substitute for the day (at least one sachet with15g PE) in an amount equivalent to their usual protein substitute PE
  Interventions: Dietary Supplement: PKU GOLIKE

INTERVENTIONS:
Dietary Supplement: PKU GOLIKE — AA protein Substitute for the dietary management of PKU, PKU GOLIKE is a food for special medicinal purposes (FSMP) for the dietary management of PKU.
  Other Names: PKU GOLIKE is a food for special medicinal purposes (FSMP) for the dietary management of PKU.

SUMMARY:
This is a 2 arm, randomised, controlled, cross-over study in 16 children with PKU. Subjects who are currently taking a Phe free/low Phe protein substitute will be recruited for a 31-day trial.

Patients will be randomised to receive:

1. The study product for 7 days as their last dose of protein substitute for the day (at least one sachet with 15g PE) in an amount equivalent to their usual protein substitute PE; or
2. An amino acid protein substitute for all daily doses for 7 days; followed by a 2-week washout period on their usual protein substitute,

and then 7 days of the other study arm.

During this time, patients/caregivers will be asked to:

* Collect 3 finger prick blood spots on days -1, 0, 6, 7, 20, 21, 27 and 28.
* Collect urine sample, second void of the day on days 0, 7, 21 and 28.
* Complete a questionnaire on sleep quality on day 0, 7, 21 and 28.
* Complete a 24 hour food diary on days -1, 0, 6, 7, 20, 21, 27 and 28.

APR will supply the study product for participants free of charge.

DETAILED DESCRIPTION:
16 children with PKU who currently take a Phe-free/low Phe protein substitute (3 or 4 doses/day) will be recruited. Subjects will replace the last daily dose of their usual protein substitute with the study product for 7 days of the 28 day trial (either days 1-7 or days 22-28 based on random allocation). On the remaining study days, subjects will take an amino acid based protein substitute for all daily doses. There will be a 2 week washout period between study arms where subjects will take their usual protein substitute. The amount of study product prescribed will be calculated to provide the same amount of protein as their usual protein substitute. The last protein substitute (PS) dose of the day (amino acids or study product) will need to be taken between 7-9pm to allow an 8-10 hour fasting period overnight. Three finger prick blood spots will be collected and analysed for phenylalanine, tyrosine and BCAA at 5am, 6am and 7am on days -1, 0, 6, 7, 20, 21, 27 and 28. For all subjects, a second void urine sample will be collected on days 0, 7, 21 and 28 for analysis of urea and creatinine. A quality of sleep questionnaire will be completed by subjects or their carers on days 0, 7, 21 and 28 and a 24 hour food diary on days -1, 0, 6, 7, 20, 21, 27 and 28. A palatability questionnaire will be completed by subjects or their carers on days 7 or 28 (at the end of the period with PKU GOLIKE, if Bars or Krunches are used). Subject visits will be on days -2 (enrolment), 0, 7, 21 and 28 where the research dietitian will collect urine samples, blood spots, questionnaires and diaries.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female PKU patients ≥5 years and ≤16 years of age.
2. Patients diagnosed with PKU via new born screening.
3. Taking a Phe free/low Phe protein substitute
4. On a low phenylalanine diet .
5. Absence of neurological deficiencies.
6. Adherence with dietary management and protein substitute.
7. Able to understand and comply with the requirements of the investigation and sign the Informed Consent Form/Assent form.

Exclusion Criteria:

1. Age <5 years old and >16 years old.
2. Patients with mild PKU or HPA.
3. On sapropterin therapy.
4. Patients with late diagnosis of PKU and neurological problems.
5. History of hypersensitivity to any excipients/components of the investigational product.
6. Pregnancy or breastfeeding during the study.
7. Any moderate to severe acute illness which in the opinion of the Investigator would interfere with the study procedures or study outcome.
8. History of poor co-operation, non-adherence with dietary management, or poor adherence to investigation procedures.
9. Participation in any other studies involving investigational or marketed products concomitantly or within two weeks prior to entry into the study.

Ages: 5 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2023-06-30 (Actual); Primary Completion 2024-05-26 (Actual); Study Completion 2024-05-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anita MacDonald, Pr., Principal Investigator — Birmingham Children's Hospital, Steelhouse Lane, Birmingham B4 6NH
Locations (1):
- Birmingham Children's Hospital Steelhouse Lane, Birmingham, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at Birmingham Hospital from June 2023 to February 2024. The first participant was enrolled on 30 June 2023 (date of informed consent signature), and the last participant was enrolled in February 2024.
Pre-assignment Details: 16 patients are recruited in the study and treated according to the study design: randomised two-periods crossover.
  3 patients are excluded from analyses due to protocol deviations. So 16 patients are included in the ITT analysis and only 13 in the PP analysis.
Groups:
- 1st PKU GOLIKE, 2nd AA Protein Substitute; 1st AA Protein Substitute 2nd PKU GOLIKE: For the study All Patients are randomised to receive:
  * The PKU GOLIKE treatment for 7 days as their last dose of protein substitute for the day in an amount equivalent to their usual protein substitute Proteine Equivalent; or
  * An amino acid protein substitute (AA treatment) for all daily doses for 7 days.
  Each the above mentioned treatments were followed by a 2-week washout period on their usual protein substitute, and then 7 days of the other study arm.
  All participants were randomized to receive both Golike and AA treatments
Period: 1st Intervention (1week)
Arm/Group | 1st PKU GOLIKE, 2nd AA Protein Substitute | 1st AA Protein Substitute 2nd PKU GOLIKE
Started | 9 | 7
Completed | 7 | 7
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0
Period: 2 Weeks Washout
Arm/Group | 1st PKU GOLIKE, 2nd AA Protein Substitute | 1st AA Protein Substitute 2nd PKU GOLIKE
Started | 9 | 7
Completed | 9 | 7
Not Completed | 0 | 0
Period: 2nd Intervention (1 Week)
Arm/Group | 1st PKU GOLIKE, 2nd AA Protein Substitute | 1st AA Protein Substitute 2nd PKU GOLIKE
Started | 9 | 7
Completed | 9 | 6
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: Sixteen patients (8 males and 8 females), included in the ITT analysis, were selected according to inclusion and exclusion criteria and randomized into the two treatment sequences in cross-over (16 patients in total)
Groups:
- All Study Participants (ITT): For the study All Patients are randomised to receive:
  * The PKU GOLIKE treatment for 7 days as their last dose of protein substitute for the day in an amount equivalent to their usual protein substitute Proteine Equivalent; or
  * An amino acid protein substitute (AA treatment) for all daily doses for 7 days.
  Each the above mentioned treatments were followed by a 2-week washout period on their usual protein substitute, and then 7 days of the other study arm.
  All participants were randomized to receive both Golike and AA treatments
Arm/Group | All Study Participants (ITT)
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.19 (3.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 14
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 16

OUTCOME MEASURES:

1. Primary Outcome: Blood Phe After 7 Days of Each Treatment
Description: Measurement of blood phenylalanine (Phe) levels
Time Frame: Mean value of Blood Sample after 7 treatment days (days 7 and 28 together depending on the period)
Population: In this cross-over study, the analysis was conducted by grouping patients data from both arms based on the type of treatment (Golike or AA) used for 7 days.
Measure: Mean (Standard Deviation); unit: µmol/L
Groups:
- All Study Participants: For the study All Patients are randomised to receive:
  * The PKU GOLIKE treatment for 7 days as their last dose of protein substitute for the day in an amount equivalent to their usual protein substitute Proteine Equivalent; or
  * An amino acid protein substitute (AA treatment) for all daily doses for 7 days.
  Each the above mentioned treatments were followed by a 2-week washout period on their usual protein substitute, and then 7 days of the other study arm.
  All participants were randomized to receive both Golike and AA treatments
Arm/Group | All Study Participants
Number analyzed (Participants) | 13
µmol/L
  Phe level Before All study partecipants from both arms start GolikeTreatment | 357.5 (155.58)
  Phe level After All study Partcipants from both arms are 7 days treated with Golike Treatment | 294.0 (149.93)
  Phe level Before All study partecipants from both arms start AA Treatment | 346.8 (143.72)
  Phe level After All study Partcipants from both arms are 7 days treated with AA Treatment | 442.4 (177.58)

2. Secondary Outcome: Dosage of Tyr in Blood (Umol/L) With Dried Blood Spots Before Breakfast
Description: Measurement of blood tyrosine (Tyr) levels
Time Frame: Mean value of Blood Sample after 7 treatment days (days 7 and 28 together depending on the period)
Measure: Mean (Standard Deviation); unit: µmol/L
Arm/Group | All Study Participants
Number analyzed (Participants) | 13
µmol/L
  Tyr level Before All study partecipants from both arms start GolikeTreatment | 46.4 (15.76)
  Tyr level after All study partecipants from both arms are 7 days treated with GolikeTreatment | 62.1 (23.43)
  Tyr level Before All study partecipants from both arms start AA Treatment | 49.5 (11.93)
  Tyr level after All study partecipants from both arms are 7 days treated with AA Treatment | 51.6 (22.02)

ADVERSE EVENTS:
Time Frame: Safety information collected from the signature of the ICF (V0) to the end of study (about 5 weeks).
Groups:
- PKU GOLIKE TREATMENT: For the study Patients are randomised to receive:
  * The PKU GOLIKE treatment for 7 days as their last dose of protein substitute for the day in an amount equivalent to their usual protein substitute Proteine Equivalent; or
  * An amino acid protein substitute (AA treatment) for all daily doses for 7 days.
  Each the above mentioned treatments were followed by a 2-week washout period on their usual protein substitute, and then 7 days of the other study arm.
  In this Arm/Group, for PKU GOLIKE treatment we consider the data of all patients after the 7 days with PKU GOLIKE as their last dose of protein substitute for the day.
- AA TREATMENT: For the study Patients are randomised to receive:
  * The PKU GOLIKE treatment for 7 days as their last dose of protein substitute for the day in an amount equivalent to their usual protein substitute Proteine Equivalent; or
  * An amino acid protein substitute (AA treatment) for all daily doses for 7 days.
  Each the above mentioned treatment were followed by a 2-week washout period on their usual protein substitute, and then 7 days of the other study arm.
  In this Arm/Group, for AA treatment we consider the data of all patients after the 7 days with AA treatment.
Arm/Group | PKU GOLIKE TREATMENT | AA TREATMENT
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 4/16 | 1/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PKU GOLIKE TREATMENT (N=16) | AA TREATMENT (N=16)
viral infections (Infections and infestations) | 2 | 1
vomiting (Infections and infestations) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The material for public dissemination will be submitted to the Sponsor for review at least sixty (60) days (or the time specified in the Protocol if longer) prior to submission for publication, public dissemination, or review by a publication committee.

All reasonable comments made by the Sponsor in relation to a proposed publication will be incorporated by the Participating Organisation and/or the Principal Investigator into the publication.

DOCUMENTS (1):
  • Study Protocol (2023-06-27): https://cdn.clinicaltrials.gov/large-docs/78/NCT05487378/Prot_000.pdf